CLINICAL TRIAL: NCT00333801
Title: The Impact of Vocational Rehabilitation on Mentally III Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4092-I; Promis Number 0052 (Other Grant/Funding Number: TVAMC); MIRB 00033 (Other: TVAMC - reference number); TVAMC 03-19 (Other: TVAMC - Year/project number); NCT00260507 (obsolete NCT alias)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic Stress Disorder; Veterans; Vocational Rehabilitation; Supported Employment; Individual Placement and Support
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vocational Rehabilitation Program (VRP) (Active Comparator): Vocational Rehabilitation Program (VRP). VRP is the treatment as usual, which mostly consisted of transitional work program (TWP) in which client is placed in a set-aside noncompetitive job for time-limited period and then pursues competitive employment at time of discharge from VRP. Limited integration with treatment team and limited follow-along supports that are time-limited
  Interventions: Behavioral: Vocational Rehabilitation Program (VRP)
- Individual Placement and Support (IPS) (Experimental): Inidividual Placement and Support (IPS). IPS Supported Employment involves an IPS specialists working with client to identify job preferences, rapidly begin community-based job search, engage in competitive employment, sustain employment via open-ended IPS follow-along supports, and integrate IPS within the PTSD treatment team.
  Interventions: Behavioral: Individual Placement and Support (IPS)

INTERVENTIONS:
Behavioral: Vocational Rehabilitation Program (VRP) — Vocational Rehabilitation Program (VRP) is a treatment-as-usual method using traditional train-place approaches, such as prevocational work skills training , compensated work therapy, or transitional work experience, which consists of temporary employment in a brokered-job with time-limited support from the VRP specialist
  Other Names: Transition work program (TWP)
  Arms: Vocational Rehabilitation Program (VRP)
Behavioral: Individual Placement and Support (IPS) — Individual Placement and Support (IPS) is an evidence--based model of supported employment that emphasizes rapid job search within client preferences, community job development, placement in a competitive job, on-the-job training, time-unlimited follow-along supports, and integration of the IPS specialist within the treatment team.
  Other Names: Supported emplooyment
  Arms: Individual Placement and Support (IPS)

SUMMARY:
To study the impact of Individual Placement and Support (IPS) supported employment (SE) compared to treatment-as-usual vocational rehabilitation program (VRP) for veterans with posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Objectives: to study the impact of Individual Placement and Support (IPS) supported employment (SE) compared to treatment-as-usual vocational rehabilitation program (VRP) for veterans with posttraumatic stress disorder (PTSD).

Research Design: This prospective randomized study evaluates the impact of IPS-SE compared to VRP on occupational, sobriety, psychiatric, and quality of life outcomes and health care costs for veterans with chronic PTSD who enter the Tuscaloosa VA Medical Center's (TVAMC) vocational rehabilitation program.

Methodology: Occupational functioning is determined primarily by whether the veteran can obtain and maintain competitive employment, and, secondarily, by time worked and wages earned for those employed. Veterans who meet inclusion criteria will be randomized to either IPS-SE or VRP. Outcomes will be assessed over a fixed 12-month observation period (beginning at randomization and computed for the entire 12-month observation period) as percent subjects employed at least one week (employed rate), and monthly employment rates (maintained employed rate). In addition, PTSD symptoms and other health-related quality of life measures will be evaluated. This strategy uses all available data during the 1-year period.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age, greater than or equal to 19 and less than 61.
* Enrollment in the TVAMC VRP
* Signed informed consent
* Chronic post-traumatic stress disorder
* Any race or ethnic origin
* Anticipation of remaining in the catchment area for the 12-month study duration

Exclusion Criteria:

* Lifetime history of severe traumatic brain injury that has resulted in severe cognitive impairment
* History of schizophrenia, schizoaffective, disorder, or bipolar I disorder
* Pending litigation
* In need of immediate detoxification.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2010-04-24 (Actual); Study Completion 2012-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lynne Davis, MD AB, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davis LL, Leon AC, Toscano R, Drebing CE, Ward LC, Parker PE, Kashner TM, Drake RE. A randomized controlled trial of supported employment among veterans with posttraumatic stress disorder. Psychiatr Serv. 2012;63(5):464-70. doi: 10.1176/appi.ps.201100340. PMID 22307881
- [Result] Davis LL, Pilkinton P, Poddar S, Blansett C, Toscano R, Parker PE. Impact of social challenges on gaining employment for veterans with posttraumatic stress disorder: an exploratory moderator analysis. Psychiatr Rehabil J. 2014 Jun;37(2):107-9. doi: 10.1037/prj0000058. Epub 2014 Apr 7. PMID 24708195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2006 to 2010 Veterans with PTSD at the Tuscaloosa VA Medical Center were enrolled in a 12-month, prospective randomized comparison of IPS Supported Employment and treatment-as-usual Vocational Rehabilitation Program (VRP).
Pre-assignment Details: 100 Veterans were enrolled; 85 were randomized to IPS-SE (n=42) or VRP (n=43) and followed 12-months. 15 participants were excluded: 2 did not have PTSD, 2 lived >100 miles away, 3 withdrew consent, 4 had exclusionary diagnosis, and 4 were not eligible to be enrolled in the VRP. Participants were allowed to continue all other treatments for PTSD.
Groups:
- Vocational Rehabilitation Program (VRP): VA Vocational Rehabilitation Program (treatment-as-usual) uses traditional train-place approaches, such as prevocational work skills training , compensated work therapy, or transitional work experience, which consists of temporary employment in a brokered-job with time-limited support from the VRP specialist
- Individual Placement and Support (IPS): Individual Placement and Support (IPS) Supported Employment (SE) emphasizes rapid job search, community job development that is keeping with participants' preferences, placement in a competitive job, on-the-job training, time-unlimited follow-along supports, and integration of IPS specialist within the treatment team.
Period: Overall Study
Arm/Group | Vocational Rehabilitation Program (VRP) | Individual Placement and Support (IPS)
Started | 43 | 42
Completed | 35 | 36
Not Completed | 8 | 6
Not completed — Moved to another state | 5 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Incarcerated | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Veterans with PTSD were randomly assigned to a treatment goup.
Groups:
- VA Vocational Rehabilitation Program (Treatment-as-usual): VA Vocational Rehabilitation Program (treatment-as-usual) uses traditional train-place approaches, such as prevocational work skills training, compensated work therapy, or transitional work experience, which consists of temporary employment in a brokered-job with time-limited support from the VRP specialist.
- Individual Placement and Support (IPS) Supported Employment: Individual Placement and Support (IPS) Supported Employment (SE) emphasizes rapid job search, community job development that is keeping with participants' preferences, placement in a competitive job, on-the-job training, time-unlimited follow-along supports, and integration of IPS specialist within the treatment team.
- Total: Total of all reporting groups
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.5) | 39.9 (11.9) | 40.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Obtain Competitive Employment
Description: The primary outcome: competitive employment (Yes or No). Competitive employment was defined as a job for regular wages in a setting that was not set aside, or sheltered, that is, the job could be held by people without a mental illness or disability and was not a set-aside job in the VRP. Day labor (babysitting, manual labor by the day, drill, temporary work for family or friends) was not considered competitive employment.
Time Frame: 1 calendar year
Population: All randomized participants were included in the analysis (intent-to-treat)
Measure: Number; unit: participants
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
participants | 12 | 32
Statistical Analysis 1: Comparison: VA Vocational Rehabilitation Program (Treatment-as-usual) vs Individual Placement and Support (IPS) Supported Employment; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: PTSD, Depression, Disability Outcomes
Description: Clinician Administered PTSD Scale for DSM-IV (CAPS) score range 0-136 with higher=more severe; Quick Inventory of Depression Scale - Clinician-rated (QIDS-CR) score range 0-27 with higher=more severe; Clinical Global Impression-Severity (CGI-S) score range 1-7 with higher=more severe; Davidson Trauma Scale (DTS) score range 0-136 with higher=more severe; and World Health Organization Disability Assessment Scale (WHODAS-II) 36-items rated on 5-point scale, from 1 (no difficulty) to 5 (extreme difficulty/cannot do) in 6 domains of life; domain scores are transformed from the total raw score (sum of items) of each domain according to the following formula: Transformed score=[(actual raw score - lowest possible raw score) / (possible raw score range)] x 100.
Time Frame: one-year
Population: All randomized participants (intent-to-treat)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
units on a scale
  CAPS | 78.4 (18.3) | 77.3 (24)
  QIDS-CR | 12.2 (4.2) | 12.3 (4.5)
  CGI-S | 5.0 (1.0) | 4.8 (0.9)
  DTS | 82.9 (28.4) | 84.9 (28.4)
  WHODAS II | 81.1 (20.5) | 82.6 (19.6)
Statistical Analysis 1: Comparison: VA Vocational Rehabilitation Program (Treatment-as-usual) vs Individual Placement and Support (IPS) Supported Employment; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Employment Outcomes (Weeks Competitively Employed)
Description: Number of weeks employed for any time in a competitive job (not set-aside job)
Time Frame: one year
Population: All randomized participants (intent-to-treat)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
weeks | 6.8 (13.8) | 21.6 (17.7)
Statistical Analysis 1: Comparison: VA Vocational Rehabilitation Program (Treatment-as-usual) vs Individual Placement and Support (IPS) Supported Employment; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Cohen's d = .93

4. Secondary Outcome: Employment Outcomes (Days Competitively Employed
Description: Number of days employed in a competitive job (not set-aside job)
Time Frame: one year
Population: All randomized participants (intent-to-treat)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
days | 29.3 (61.9) | 83.8 (80.6)

5. Secondary Outcome: Employment Outcomes (Hours Competitively Employed)
Description: hours employed in a competitive (not set-aside) job
Time Frame: one year
Population: All randomized participants (intent-to-treat)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
hours | 236 (494) | 656 (661)

6. Secondary Outcome: Employment Outcomes (Gross Income Competitive)
Description: total gross income (US dollars) from all competitive wages, salary, commissions
Time Frame: one year
Population: All randomized participants (intent-to-treat)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
US dollars | 2,601 (6,009) | 9,264 (13,294)

7. Secondary Outcome: Employment Outcomes (Total Gross Income From All Sources
Description: total gross income from all sources of work including noncompetitive and competitive jobs
Time Frame: one year
Population: All randomized participants (intent-to-treat)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Number analyzed (Participants) | 43 | 42
US dollars | 3,909 (6,212) | 13,449 (9,308)

ADVERSE EVENTS:
Time Frame: Serious adverse events were carefully reviewed with the patients during their participation in the study (1 year), regardless of cause. All serious adverse events were reported to the IRB within 48 hours from the time the PI learned of the event.
Arm/Group | VA Vocational Rehabilitation Program (Treatment-as-usual) | Individual Placement and Support (IPS) Supported Employment
Serious Adverse Events (participants affected / at risk) | 11/43 | 5/42
Other Adverse Events (participants affected / at risk) | 7/43 | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VA Vocational Rehabilitation Program (Treatment-as-usual) (N=43) | Individual Placement and Support (IPS) Supported Employment (N=42)
Suicidal Ideation (Psychiatric disorders) | 5 | 4
Severe Staph Infection (Infections and infestations) | 1 | 0
Surgical procedure (Surgical and medical procedures) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Motor Vehicle Accident complications (General disorders) | 1 | 0
Medical Stabilization (General disorders) | 1 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abnormally high blood pressure (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VA Vocational Rehabilitation Program (Treatment-as-usual) (N=43) | Individual Placement and Support (IPS) Supported Employment (N=42)
Severe migraine headache (General disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Injury to finger (Injury, poisoning and procedural complications) | 1 | 0
Hypertrophy adnoids (Ear and labyrinth disorders) | 0 | 1
Neck swelling (General disorders) | 1 | 0
Alcohol withdrawal (Injury, poisoning and procedural complications) | 2 | 0
Cyst underarm (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
The elements of the study that limit generalizability include the single-site design, the small number of IPS interventionists, low number of women in the sample, and the exclusion of nonveterans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes